CLINICAL TRIAL: NCT05387330
Title: Monitoring of Soluble L-selectin (sCD62L) and Secreted Protein Acidic Rich in Cysteine in Chronic Myeloid Leukemia Patients Treated by Imatinib
Brief Title: Dynamic Changes in the Levels of sCD62L and SPARC in Chronic Myeloid Leukemia Patients During Imatinib Treatment
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohamed Elkholy, Instructor of Clinical Pharmacy, Tanta University
Other Study IDs: 9093595
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Soluble L-selectin, sCD62L, SPARC, Imatinib, CML
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and serum blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CP-CML patients: Twenty five newly diagnosed CP-CML patients. Plasma sCD62L and serum SPARC levels were measured using commercially available ELISA kits
  Interventions: Diagnostic Test: ELISA kit
- Control: Ten matched controls were enrolled. Plasma sCD62L and serum SPARC levels were measured using commercially available ELISA kits
  Interventions: Diagnostic Test: ELISA kit

INTERVENTIONS:
Diagnostic Test: ELISA kit — Sandwich ELISA kit for the accurate quantitative detection of sCD62L and SPARC in human plasma and serum samples.

SUMMARY:
This study aims to monitor the levels of soluble L-selectin (sCD62L) and secreted protein acidic rich in cysteine (SPARC) in chronic phase chronic myeloid leukemia (CP-CML) patients at baseline and after three and six months of imatinib therapy and evaluated the effect of imatinib on their levels and correlated their levels to clinical and laboratory parameters.

DETAILED DESCRIPTION:
Chronic myelogenous leukemia (CML) is a clonal myeloproliferative disorder characterized by the reciprocal t (9:22) chromosomal translocation. This rearrangement produces abnormal chromosome called Philadelphia chromosome carrying the chimeric BCR-ABL oncoprotein which encodes for tyrosine kinase (TK). The Break Point Cluster Region- Abelson (BCR-ABL) fusion oncoprotein activates the various downstream signaling pathways causing reduced hematopoietic cell differentiation, decreased apoptosis, enhance proliferation and survival of leukemic cells. CML remains incurable for the most part, and only allogeneic hematopoietic stem cell transplantation can eradicate and cure CML. This is probably because quiescent leukemic stem cells are resistant to tyrosine kinase inhibitors (TKIs).

Imatinib (IM) was the first tyrosine kinase inhibitor to receive approval by the Food and Drug Administration for the treatment of patients with CML-CP. It acts via competitive inhibition at the ATP - binding site of the BCR-ABL protein, which results in the inhibition of phosphorylation of proteins involved in signal transduction. It inhibits the BCR-ABL kinase.

L-selectin is a glycoprotein which is one of three members in a family of cell adhesion molecules called selectins. L-selectin is expressed on most leukocytes and it appears to play an important role in the early stages of leukocyte-endothelial cell interaction. L-selectin is a critical molecule for the leukocyte-endothelial cell interaction that results in migration of naïve T-cells into peripheral lymph nodes and inflammatory locales such as: tumor microenvironment.

Secreted Protein, Acidic Rich in Cysteine (SPARC) is a multi-functional matricellular glycoprotein with growth inhibitory and anti-angiogenic activity in some cell types. This protein has counter adhesive properties, has effects on cell shape, immune surveillance, angiogenesis and inhibits cell proliferation. SPARC is multifunctional calcium binding matricellular glycoprotein, participates in tissue remodeling, morphogenesis and bone mineralization and is secreted by different types of cells such as: osteoblasts, fibroblasts and endothelial cells. SPARC binds Vascular Endothelial Growth Factor (VEGF), preventing VEGF induced tyrosine phosphorylation of VEGFR1 and antagonizing its pro-angiogenic effects. The role of SPARC in tumor genesis appears to be cell-type specific due to its diverse function in given microenvironment.

sCD62L and SPARC analyzed using commercially available ELISA kit.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes.
* Newly diagnosed patient with chronic phase, Philadelphia chromosome positive (Ph+) CML.
* Age ≥ 18 years.

Exclusion Criteria:

* Patients in blastic or accelerated phase of chronic myeloid leukemia.
* Previous treatment with Imatinib.
* Pregnancy and lactation.
* Severe hepatic dysfunction.
* Kidney dysfunction.
* Intolerant or incompliant to imatinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed CP-CML patients were invited to be enrolled in this study. Patients were diagnosed according to ELN guidelines. Full patient history taken and proper information sheets completed for all participants.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-07-25 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Dynamic changes of sCD62L and SPARC levels in CP-CML patients during imatinib treatment | Baseline and after three and six months of treatment
  Monitoring the changes in sCD62L and SPARC levels at baseline and after three and six months of imatinib treatment

SECONDARY OUTCOMES:
Correlations of sCD62L or SPARC levels with laboratory and clinical parameters | Baseline and after three and six months of treatment
  Correlations of sCD62L or SPARC levels with BCR-ABL1%, sokal risk score, spleen size, age and white blood cells, neutrophils, monocytes and lymphocytes counts at baseline and after three and six months of imatinib treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud M Elkholy, Bachelor, Principal Investigator — Clinical Pharmacy Department, Faculty of Pharmacy, Al Salam University in Egypt; Sahar M El-Haggar, Ph D, Principal Investigator — Clinical Pharmacy Department, Faculty of Pharmacy, Tanta University; Maryan W Fahmi, Ph D, Principal Investigator — Medical oncology unit, Internal medicine Department, Faculty of medicine
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sonoyama J, Matsumura I, Ezoe S, Satoh Y, Zhang X, Kataoka Y, Takai E, Mizuki M, Machii T, Wakao H, Kanakura Y. Functional cooperation among Ras, STAT5, and phosphatidylinositol 3-kinase is required for full oncogenic activities of BCR/ABL in K562 cells. J Biol Chem. 2002 Mar 8;277(10):8076-82. doi: 10.1074/jbc.M111501200. Epub 2002 Jan 4. PMID 11779872
- [Background] Krause DS, Lazarides K, Lewis JB, von Andrian UH, Van Etten RA. Selectins and their ligands are required for homing and engraftment of BCR-ABL1+ leukemic stem cells in the bone marrow niche. Blood. 2014 Feb 27;123(9):1361-71. doi: 10.1182/blood-2013-11-538694. Epub 2014 Jan 6. PMID 24394666
- [Background] Sopper S, Mustjoki S, White D, Hughes T, Valent P, Burchert A, Gjertsen BT, Gastl G, Baldauf M, Trajanoski Z, Giles F, Hochhaus A, Ernst T, Schenk T, Janssen JJ, Ossenkoppele GJ, Porkka K, Wolf D. Reduced CD62L Expression on T Cells and Increased Soluble CD62L Levels Predict Molecular Response to Tyrosine Kinase Inhibitor Therapy in Early Chronic-Phase Chronic Myelogenous Leukemia. J Clin Oncol. 2017 Jan 10;35(2):175-184. doi: 10.1200/JCO.2016.67.0893. Epub 2016 Nov 7. PMID 28056193
- [Background] Podhajcer OL, Benedetti L, Girotti MR, Prada F, Salvatierra E, Llera AS. The role of the matricellular protein SPARC in the dynamic interaction between the tumor and the host. Cancer Metastasis Rev. 2008 Sep;27(3):523-37. doi: 10.1007/s10555-008-9135-x. PMID 18459035